CLINICAL TRIAL: NCT02684214
Title: Implementing Prevention Plus for Childhood Overweight and Obesity in Food Secure and Insecure Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Collaborators: Cherokee Health Systems (Unknown); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Hollie Raynor, Professor, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UTK IRB-15-02680-FB
Record Dates: First submitted 2016-02-02; First posted 2016-02-17 (Estimated); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Obesity; Childhood Obesity
Keywords: food security
MeSH Terms: conditions — Obesity; Pediatric Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Food secure families (Experimental): high and marginal household food security
  Interventions: Behavioral: Prevention Plus +; Behavioral: Prevention Plus -
- Food insecure families (Experimental): low and very low household food security
  Interventions: Behavioral: Prevention Plus +; Behavioral: Prevention Plus -

INTERVENTIONS:
Behavioral: Prevention Plus + — Families will receive 6 monthly newsletters and meet with a BHC at the clinic for 30 minutes during months 1, 3, and 5. Child height and weight will be taken. Families will receive feedback about growth and the weight status of their child. The session materials will be reviewed and behavioral parenting strategies will be encouraged to aid with changing two dietary and two leisure-time activity (energy balance) behaviors of the child. The caretaker will also change the same energy balance behaviors as the child, as adult caretakers can then model healthy behaviors. The caretaker and child will be encouraged to change and self-monitor energy balance behaviors with the use of the picture-based diaries. During months 2, 4, and 6, BHCs will complete a 20-minute phone call with the caretaker. Caretakers will be asked to measure the height and weight of their child, calculate BMI and plot it on the BMI-for-age growth chart prior to the call. The BHC will provide feedback.
Behavioral: Prevention Plus - — This condition will be identical to PP+ except that caretakers will not receive any energy balance behavior goals. Additionally, the caretaker will not self-monitor energy balance behaviors. The focus will be on all other behavioral parenting strategies to assist the child with making changes in the targeted behaviors.

SUMMARY:
The ability of Prevention Plus to improve weight status when delivered by primary care providers is unknown, and the influence of household food security status as a moderator in the treatment of childhood obesity has never been examined. Thus, the investigators will conduct a randomized trial examining Prevention Plus delivered by CHS primary care providers on child zBMI in underserved children receiving their primary care at CHS who are overweight and obese, and test the moderating effect of household food security status on Prevention Plus delivered with and without caretaker goals

DETAILED DESCRIPTION:
Intervention

PP+

Following baseline assessment, children will continue to receive standard care at CHS and the monthly newsletter. Additionally, each family will be provided with a scale; wall growth chart to measure height; a BMI wheel to calculate BMI; a BMI-for-age growth chart; a binder for intervention materials; a self-monitoring diary to record child's monthly height, weight, BMI and BMI percentile; and picture-based diaries to monitor daily energy balance behaviors. Family materials provided at each session will outline a process to measure growth and include information about how children grow, as well as cover behavioral parenting strategies to assist with changing child behavior for energy balance behaviors.

Families will meet in person with a BHC at the CHS clinic in which they receive care for 30 minutes during months 1, 3, and 5. In these sessions, child height and weight will be taken, and BMI will be plotted on the BMI-for-age growth chart. Families will receive feedback about growth and the weight status of their child. Additionally, the session materials will be reviewed and behavioral parenting strategies will be encouraged to aid with changing two dietary and two leisure-time activity (energy balance) behaviors of the child. As is traditional in a family-based approach, the caretaker will also change the same energy balance behaviors as the child, as adult caretakers can then model healthy behaviors for the child, assisting the child in learning the new weight-related behaviors.13 Thus, both the caretaker and child will be encouraged to change and self-monitor energy balance behaviors with the use of the picture-based diaries.

During months 2, 4, and 6, BHCs will complete a 20-minute phone call with the caretaker. Caretakers will be asked to measure the height and weight of their child, calculate BMI and plot it on the BMI-for-age growth chart prior to the call. During the call, the BHC will provide feedback on the changes in child growth since the previous contact. Additionally, the BHC will discuss the family's progress on achieving child and caretaker energy balance behavior goals and implementation of behavioral parenting strategies.

The child's energy balance behavioral goals will be to consume < 3 sugar-sweetened beverage (e.g., regular carbonated soft drinks, sports drinks, lemonades, ice teas, flavored milk, juice drinks < 100% juice, and punches) servings /wk, ≥1 ½ cups/day of whole vegetables and ≥ 1 cup/day of whole fruit, engage in ≥ 60 minutes/day of moderate- to vigorous-intensity physical activity, and reduce TV viewing to < 2 hours/day. The caretaker's energy balance behavioral goals will be to consume < 3 sugar-sweetened beverage servings/wk, ≥ 2 ½ cups/day of whole vegetables and ≥ 1 ½ cups/day of whole fruit, engage in ≥ 150 minutes of moderate- to vigorous-intensity physical activity per week, and reduce TV viewing to < 10 hours/wk. To increase self-efficacy, the goals will be incrementally increased, with families implementing the full program goals at month four. Additionally, children and caretakers will be asked to achieve at least three of the five goals each day (child) or week (adult caretaker).

PP-

This condition will be identical to PP+ except that caretakers will not receive any energy balance behavior goals. Additionally, the caretaker will not self-monitor energy balance behaviors. The focus will be on all other behavioral parenting strategies to assist the child with making changes in the targeted behaviors (i.e., stimulus control, positive reinforcement, and assisting child in self-monitoring energy-balance behaviors).

ELIGIBILITY:
Inclusion Criteria:

* patient at five clinics (Alcoa [Blount County], Knox County Pediatrics [Knox County], Maynardville [Union County], Seymour [Sevier County], and Talbott [Hamblen County]).
* BMI > 85th percentile
* have an adult (> 18 years) female caretaker living in the household willing to participate in the program.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2016-04; Primary Completion 2018-12-31 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Target Population Denominator | 2 years
  CHS' Electronic Health Record will allow the number of children meeting eligibility criteria to be determined and the target population denominator identified.
Basic demographic information and weight history | Baseline
  Basic demographic information (e.g., child's gender and age; parent's, gender, age, and education level) and health history will be obtained at baseline.
Household Food Security Status assessed with the Household Food Security Module | Baseline
  This module consists of three stages of adult-referenced questions and two stages of child-referenced questions. The time frame that will be used to assess household food security status will be in the previous 30 days (the module is validated for a 12-month or 30 day time frame). Families will be scored as food secure (high and marginal household food security) or food insecure (low and very low household food security). This will be administered at 0 and 6 months (to assess if household food security status changed during the intervention).
z-BMI | Change from baseline to 6-months
Child and caretaker dietary intake be assessed via 3-day food diaries | Change from baseline to 6 months
  During the 3-day period(1 weekend day, 2 weekdays), if the child is under the supervision/care of another adult other than the caretaker, the caretaker will be instructed to obtain information from this other adult about what the child consumed. Families will be provided with measuring cups and spoons and two-dimensional aids to help with accuracy of recording. Caretakers will be trained on how to complete the food diaries. Diaries will be reviewed to ensure that information about food consumption is complete. Nutrition data will be analyzed using the Nutrition Data System Research Software (NDSR)
Activity assessed via Previous Day Physical Activity Recall | Change from baseline to 6 months
  This is a self-report questionnaire that assesses all activity, both physical activity and sedentary behavior, in children and adolescents. Specifically, the PD-PAR collects information on screen time, allowing measurement of this targeted behavior. This questionnaire will be completed at 0 and 6 by both children and caretakers. The compendium of physical activities for youth will be used to estimate energy expenditure from the PD-PAR. Dependent variables will be minutes of physical activity and screen time, percent of time spent in sedentary behavior and moderate- to vigorous-intensity physical activity, and overall daily metabolic equivalent (MET) value.
Quality Control | 2 years
Parent Weight History | baseline
  parent weight loss history will be obtained via a questionnaire

SECONDARY OUTCOMES:
Participation Rate | 2 years
Participant vs. non-participant Characteristics | 2 years
  The Electronic Health Record (EHR) will allow comparisons on demographic and health characteristics between eligible children who participate vs. those who do not. CHS IT staff will extract these data from the EHR during the last 4 months of the project.
Program Adherence assessed with a a behavioral checklist | 2 years
  Adherence to delivery of intervention for each session will be ascertained using a behavioral checklist
Intervention Fidelity assessed with a behavioral checkllist | 2 years
  Fidelity will be ascertained by discussion of parent goals regarding energy balance behaviors in PP+ and lack of discussion regarding parent goals or changing energy balance behaviors in PP- and/or refocusing session on behavioral parenting strategies as needed.
program sustainability assessed via interviews | 2 years
  Individual interviews will be conducted with at least 2 providers from each participating CHS clinic and all BHCs who delivered the PP programs to ascertain satisfaction with the approach and perceptions of sustainability of the intervention in CHS. It is anticipated that 10 CHS staff and 2 BHCs will be recruited for the 30 minute interview.
  Dr. Barroso will lead this process. Interview scripts will be developed via an iterative process involving the research team.

CONTACTS AND LOCATIONS:
Locations (1):
- Healthy Eating and Activity Laboratory, University of Tennessee, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kranz S, Mitchell DC, Smiciklas-Wright H, Huang SH, Kumanyika SK, Stettler N. Consumption of recommended food groups among children from medically underserved communities. J Am Diet Assoc. 2009 Apr;109(4):702-7. doi: 10.1016/j.jada.2008.12.018. PMID 19328266
- [Background] Nackers LM, Appelhans BM. Food insecurity is linked to a food environment promoting obesity in households with children. J Nutr Educ Behav. 2013 Nov-Dec;45(6):780-4. doi: 10.1016/j.jneb.2013.08.001. Epub 2013 Sep 8. PMID 24021456
- [Background] Spear BA, Barlow SE, Ervin C, Ludwig DS, Saelens BE, Schetzina KE, Taveras EM. Recommendations for treatment of child and adolescent overweight and obesity. Pediatrics. 2007 Dec;120 Suppl 4:S254-88. doi: 10.1542/peds.2007-2329F. PMID 18055654
- [Background] Raynor HA, Osterholt KM, Hart CN, Jelalian E, Vivier P, Wing RR. Efficacy of U.S. paediatric obesity primary care guidelines: two randomized trials. Pediatr Obes. 2012 Feb;7(1):28-38. doi: 10.1111/j.2047-6310.2011.00005.x. Epub 2011 Dec 13. PMID 22434737
- [Background] Looney SM, Raynor HA. Examining the effect of three low-intensity pediatric obesity interventions: a pilot randomized controlled trial. Clin Pediatr (Phila). 2014 Dec;53(14):1367-74. doi: 10.1177/0009922814541803. Epub 2014 Jul 7. PMID 25006118
- [Background] Kitzman-Ulrich H, Wilson DK, St George SM, Lawman H, Segal M, Fairchild A. The integration of a family systems approach for understanding youth obesity, physical activity, and dietary programs. Clin Child Fam Psychol Rev. 2010 Sep;13(3):231-53. doi: 10.1007/s10567-010-0073-0. PMID 20689989
- [Background] Janicke DM, Sallinen BJ, Perri MG, Lutes LD, Huerta M, Silverstein JH, Brumback B. Comparison of parent-only vs family-based interventions for overweight children in underserved rural settings: outcomes from project STORY. Arch Pediatr Adolesc Med. 2008 Dec;162(12):1119-25. doi: 10.1001/archpedi.162.12.1119. PMID 19047538
- [Background] Wright JA, Phillips BD, Watson BL, Newby PK, Norman GJ, Adams WG. Randomized trial of a family-based, automated, conversational obesity treatment program for underserved populations. Obesity (Silver Spring). 2013 Sep;21(9):E369-78. doi: 10.1002/oby.20388. Epub 2013 Jun 11. PMID 23512915
- [Background] Dinour LM, Bergen D, Yeh MC. The food insecurity-obesity paradox: a review of the literature and the role food stamps may play. J Am Diet Assoc. 2007 Nov;107(11):1952-61. doi: 10.1016/j.jada.2007.08.006. PMID 17964316
- [Background] Metallinos-Katsaras E, Must A, Gorman K. A longitudinal study of food insecurity on obesity in preschool children. J Acad Nutr Diet. 2012 Dec;112(12):1949-58. doi: 10.1016/j.jand.2012.08.031. PMID 23174682
- [Background] Martin MA, Lippert AM. Feeding her children, but risking her health: the intersection of gender, household food insecurity and obesity. Soc Sci Med. 2012 Jun;74(11):1754-64. doi: 10.1016/j.socscimed.2011.11.013. Epub 2011 Dec 20. PMID 22245381
- [Background] Skelton JA, Buehler C, Irby MB, Grzywacz JG. Where are family theories in family-based obesity treatment?: conceptualizing the study of families in pediatric weight management. Int J Obes (Lond). 2012 Jul;36(7):891-900. doi: 10.1038/ijo.2012.56. Epub 2012 Apr 24. PMID 22531090
- [Background] Akers JD, Estabrooks PA, Davy BM. Translational research: bridging the gap between long-term weight loss maintenance research and practice. J Am Diet Assoc. 2010 Oct;110(10):1511-22, 1522.e1-3. doi: 10.1016/j.jada.2010.07.005. PMID 20869490
- [Background] Glasgow RE, Klesges LM, Dzewaltowski DA, Bull SS, Estabrooks P. The future of health behavior change research: what is needed to improve translation of research into health promotion practice? Ann Behav Med. 2004 Feb;27(1):3-12. doi: 10.1207/s15324796abm2701_2. PMID 14979858
- [Background] Livingstone MB, Robson PJ, Wallace JM. Issues in dietary intake assessment of children and adolescents. Br J Nutr. 2004 Oct;92 Suppl 2:S213-22. doi: 10.1079/bjn20041169. PMID 15522159
- [Background] Livingstone MB, Robson PJ. Measurement of dietary intake in children. Proc Nutr Soc. 2000 May;59(2):279-93. doi: 10.1017/s0029665100000318. PMID 10946797
- [Background] Guenther PM, Casavale KO, Reedy J, Kirkpatrick SI, Hiza HA, Kuczynski KJ, Kahle LL, Krebs-Smith SM. Update of the Healthy Eating Index: HEI-2010. J Acad Nutr Diet. 2013 Apr;113(4):569-80. doi: 10.1016/j.jand.2012.12.016. Epub 2013 Feb 13. PMID 23415502
- [Background] Weston AT, Petosa R, Pate RR. Validation of an instrument for measurement of physical activity in youth. Med Sci Sports Exerc. 1997 Jan;29(1):138-43. doi: 10.1097/00005768-199701000-00020. PMID 9000167
- [Background] Ridley K, Ainsworth BE, Olds TS. Development of a compendium of energy expenditures for youth. Int J Behav Nutr Phys Act. 2008 Sep 10;5:45. doi: 10.1186/1479-5868-5-45. PMID 18782458